CLINICAL TRIAL: NCT06820645
Title: CALM: Calcium Administration in Life-saving Management of Trauma Patients Undergoing Massive Hemorrhage Protocol: a Single Centre Feasibility Study
Brief Title: Calcium Administration in Life-saving Management During Massive Hemorrhage
Acronym: CALM
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Ian Ball, Associate Professor, Department of Medicine, London Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 15231
Record Dates: First submitted 2025-01-13; First posted 2025-02-11 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-01

CONDITIONS: Massive Hemorrhage; Trauma; Hypocalcemia
Keywords: Calcium; Massive Hemorrhage Protocol
MeSH Terms: conditions — Wounds and Injuries; Hypocalcemia | interventions — Calcium Gluconate; Calcium; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Calcium Receiving (Experimental): Patients will receive standard care according to the Ontario MHP with calcium gluconate administration after every 4 units of RBCs given during the MHP.
  Interventions: Drug: calcium gluconate
- Placebo Comparator (Placebo Comparator): Patients will receive standard care according to the Ontario MHP with saline placebo administration after every 4 units of RBCs given during the MHP.
  Interventions: Drug: Control: Placebo

INTERVENTIONS:
Drug: calcium gluconate — 3g IV or IO calcium gluconate.
  Other Names: Calcium
  Arms: Calcium Receiving
Drug: Control: Placebo — 3g of IV or IO saline placebo.
  Other Names: saline
  Arms: Placebo Comparator

SUMMARY:
This study evaluates the feasibility of conducting a larger study on the impact of treating massive hemorrhage with calcium in trauma patients. Patients undergoing the Massive Hemorrhage Protocol (MHP) will be randomly assigned to receive either calcium gluconate or placebo drug after every 4 packs of units of RBCs received during the MHP.

DETAILED DESCRIPTION:
The treatment of hemorrhage with blood products has been well studied, however very little literature exists on the administration of specific electrolytes such as calcium. Citrate is added to blood products to prevent coagulation by chelating free calcium. This process reduces serum calcium and can lead to hypocalcemia, especially in trauma patients who have altered metabolism, hypovolemia, and receive large quantities of blood products. The majority of trauma patients have hypocalcemia upon arrival at the hospital. Serum hypocalcemia in trauma patients matters because calcium is crucial for bleeding control due to its contributions to platelet function, coagulation, and vasoconstriction. Calcium is also essential for other physiological functions during trauma, such as heart and smooth muscle contractility. It is likely due to these key roles that the literature demonstrates hypocalcemia's association with increased mortality, bleeding, blood transfusion requirements, and coagulopathy.

The primary objective of our proposed trial is to assess the feasibility of conducting an interventional calcium trial on patients undergoing the Massive Hemorrhage Protocol (MHP). Feasibility will be evaluated through the recruitment of patients, adherence to protocol, as well as assessment of any protocol violations that occur during the trial. Secondary objectives of our trial include analyzing the effect calcium supplementation has on patient ionized calcium (iCa) level, total blood product transfused, hemodynamic instability, ICU mortality, and hospital mortality.

The investigators will complete a single-centre, double-blinded randomized control feasibility trial. Both trial arms will receive study drug in accordance with Ontario's Massive Hemorrhage Protocol (MHP). After every 4 units of RBCs, the treatment group will receive 3g of calcium gluconate and the control arm will receive saline placebo. Results will be assessed for feasibility to inform the development of a larger trial.

ELIGIBILITY:
Inclusion Criteria:

* Adult trauma patients undergoing the MHP at Victoria Hospital, London, Ontario

Exclusion Criteria:

* Under the age of 18
* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Feasibility | Through study completion, an estimate of 1 year
  Recruitment of patients, adherence to the protocol, and assessment of any protocol violations that occur during the trial.

SECONDARY OUTCOMES:
Ionized calcium (iCa) | An estimate of up to 24 hours
  Change in iCa between first iCa measurement during MHP and first iCa measurement after MHP
Total blood product transfused | Duration of MHP, an average of 1 hour
  Number and type of blood products transfused during the MHP
Hemodynamic instability | Duration of MHP, an average of 1 hour
  Mean blood pressure during the MHP
ICU mortality | 30 days
Hospital mortality | 30 days

REFERENCES:
- [Background] Imamoto T, Sawano M. Effect of ionized calcium level on short-term prognosis in severe multiple trauma patients: a clinical study. Trauma Surg Acute Care Open. 2023 Jun 30;8(1):e001083. doi: 10.1136/tsaco-2022-001083. eCollection 2023. PMID 37396952
- [Background] Morotti A, Charidimou A, Phuah CL, Jessel MJ, Schwab K, Ayres AM, Romero JM, Viswanathan A, Gurol ME, Greenberg SM, Anderson CD, Rosand J, Goldstein JN. Association Between Serum Calcium Level and Extent of Bleeding in Patients With Intracerebral Hemorrhage. JAMA Neurol. 2016 Nov 1;73(11):1285-1290. doi: 10.1001/jamaneurol.2016.2252. PMID 27598746
- [Background] Kronstedt S, Roberts N, Ditzel R, Elder J, Steen A, Thompson K, Anderson J, Siegler J. Hypocalcemia as a predictor of mortality and transfusion. A scoping review of hypocalcemia in trauma and hemostatic resuscitation. Transfusion. 2022 Aug;62 Suppl 1(Suppl 1):S158-S166. doi: 10.1111/trf.16965. Epub 2022 Jun 24. PMID 35748676
- [Background] Vasudeva M, Mathew JK, Groombridge C, Tee JW, Johnny CS, Maini A, Fitzgerald MC. Hypocalcemia in trauma patients: A systematic review. J Trauma Acute Care Surg. 2021 Feb 1;90(2):396-402. doi: 10.1097/TA.0000000000003027. PMID 33196630
- [Background] Vincent JL, Bredas P, Jankowski S, Kahn RJ. Correction of hypocalcaemia in the critically ill: what is the haemodynamic benefit? Intensive Care Med. 1995 Oct;21(10):838-41. doi: 10.1007/BF01700968. PMID 8557873
- [Background] Giancarelli A, Birrer KL, Alban RF, Hobbs BP, Liu-DeRyke X. Hypocalcemia in trauma patients receiving massive transfusion. J Surg Res. 2016 May 1;202(1):182-7. doi: 10.1016/j.jss.2015.12.036. Epub 2015 Dec 30. PMID 27083965
- [Background] Bell KT, Salmon CM, Purdy BA, Canfield SG. EVALUATION OF TRANEXAMIC ACID AND CALCIUM CHLORIDE IN MAJOR TRAUMAS IN A PREHOSPITAL SETTING: A NARRATIVE REVIEW. Shock. 2023 Sep 1;60(3):325-332. doi: 10.1097/SHK.0000000000002177. Epub 2023 Jul 12. PMID 37477447
- [Background] Torres CM, Kenzik KM, Saillant NN, Scantling DR, Sanchez SE, Brahmbhatt TS, Dechert TA, Sakran JV. Timing to First Whole Blood Transfusion and Survival Following Severe Hemorrhage in Trauma Patients. JAMA Surg. 2024 Apr 1;159(4):374-381. doi: 10.1001/jamasurg.2023.7178. PMID 38294820
- [Background] Borgman MA, Spinella PC, Perkins JG, Grathwohl KW, Repine T, Beekley AC, Sebesta J, Jenkins D, Wade CE, Holcomb JB. The ratio of blood products transfused affects mortality in patients receiving massive transfusions at a combat support hospital. J Trauma. 2007 Oct;63(4):805-13. doi: 10.1097/TA.0b013e3181271ba3. PMID 18090009
- [Background] Holcomb JB, Tilley BC, Baraniuk S, Fox EE, Wade CE, Podbielski JM, del Junco DJ, Brasel KJ, Bulger EM, Callcut RA, Cohen MJ, Cotton BA, Fabian TC, Inaba K, Kerby JD, Muskat P, O'Keeffe T, Rizoli S, Robinson BR, Scalea TM, Schreiber MA, Stein DM, Weinberg JA, Callum JL, Hess JR, Matijevic N, Miller CN, Pittet JF, Hoyt DB, Pearson GD, Leroux B, van Belle G; PROPPR Study Group. Transfusion of plasma, platelets, and red blood cells in a 1:1:1 vs a 1:1:2 ratio and mortality in patients with severe trauma: the PROPPR randomized clinical trial. JAMA. 2015 Feb 3;313(5):471-82. doi: 10.1001/jama.2015.12. PMID 25647203
- [Background] Saviano A, Perotti C, Zanza C, Longhitano Y, Ojetti V, Franceschi F, Bellou A, Piccioni A, Jannelli E, Ceresa IF, Savioli G. Blood Transfusion for Major Trauma in Emergency Department. Diagnostics (Basel). 2024 Mar 27;14(7):708. doi: 10.3390/diagnostics14070708. PMID 38611621